CLINICAL TRIAL: NCT06079762
Title: AGE SELF CARE: Promoting Healthy Aging Through a Group Visit Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Julia Loewenthal, Principal Investigator, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023P001407
Record Dates: First submitted 2023-09-29; First posted 2023-10-12 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Frailty; Aging; Frailty Syndrome; Frail Elderly Syndrome
Keywords: yoga; mind-body; pre-frail; healthy aging
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: single-group feasibility/acceptability, stage I (NIH stage model for behavioral intervention development)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AGE SELF CARE group visit program (Experimental): Participants will take part in 8 weekly 90-minute virtual group visit program sessions
  Interventions: Behavioral: AGE SELF CARE group visit program

INTERVENTIONS:
Behavioral: AGE SELF CARE group visit program — AGE SELF CARE: "Adaptation, Growth, and Engagement; Socialization, Empowerment, Learning, and Function; and Community Activation for Resilience in Elderhood," is a virtual group visit program. It includes education and behavioral change elements in the broad areas of self/health, home environment, and community. There are 8 weekly 90-minute virtual sessions facilitated by an aging expert (e.g., geriatrician). Examples of topics include "Aging Well: The Power of Movement," "People Can Change, Homes Can Too," and "Social World."

SUMMARY:
Aim 1: To assess the feasibility and acceptability of delivering AGE SELF CARE through virtual medical group visits by measuring recruitment rate, adherence, and participant satisfaction.

Hypothesis 1: It will be feasible to recruit 12 older adults who are pre-frail. Hypothesis 2: At least 70% of participants will attend 6 of 8 group visit sessions.

Hypothesis 3: At least 70% of participants will report satisfaction with the program.

Aim 2: Determine the feasibility and burden of measuring frailty in this study by different instruments.

Hypothesis 1: At least 70% of participants will complete portions of all frailty assessments.

Hypothesis 2: Participants will not find testing to be burdensome and measures may be completed in 60 minutes or less.

Hypothesis 3: Mean gait speed and frailty index will improve from baseline to post-intervention.

DETAILED DESCRIPTION:
Study Design: pilot study

Setting: BWH Osher Clinical Center for Integrative Medicine, or "OCC", is a collaboration between BWH and Harvard Medical School (HMS), focused on enhancing human health, resilience, and quality of life through translational research, clinical practice, and education in integrative medicine. The OCC is comprised of an interdisciplinary team of physicians, chiropractors, acupuncturists, massage therapists, coaches, nutritionists, craniosacral therapists, and other practitioners who treat patients with a variety of conditions. Patients across New England regularly access the OCC through self-referral or referral from primary care or subspecialty practices.

Participants: Community-dwelling adults aged 65 years and older who are pre-frail (based on FRAIL) during the initial study visit (n=12).

Intervention: AGE SELF CARE consists of 8 weekly 90-minute virtual group visits, with approximately 12 participants in each group. Sessions focus on chronic disease management; healthy lifestyle education, including nutrition, physical activity, sleep, stress management, and socialization; home adaptation to optimize the home environment for usability and safety with aging; and anticipatory guidance. Educational materials include a library of handouts and pre-recorded videos from interdisciplinary team members about a topic. The group applies learning to their own lives, develops personal goals, and reports back about brief home activities or practices.

Sessions will be modified and targeted toward frailty prevention according to existing data and published guidelines. For example, the Mediterranean diet will be discussed as a nutritional approach that can reduce frailty progression. Physical activity guidelines will focus on resistance training to simulate daily activities, power training, balance exercise, and mind-body movement. Finally, sessions will include information on home safety modification and polypharmacy.

ELIGIBILITY:
Inclusion criteria:

1. Community-dwelling adults age 65+.
2. Pre-frail (1-2 points on FRAIL scale) during pre-screening.
3. Agree to participate and commit to all study procedures.
4. Able to speak English.
5. Access to and ability to use a smartphone, tablet, or computer and broadband internet.

Exclusion criteria:

1. Younger than age 65.
2. Robust (0 points) or frail (3+ points) on FRAIL scale during phone screening.
3. Established diagnosis of dementia.
4. Untreated psychiatric symptoms affecting group participation.
5. Hearing or visual impairment affecting participation in a virtual program.

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | Baseline
  Proportion of contacted potential participants who enrolled in the study
Completion of testing | Baseline and immediately after the intervention
  Proportion of enrolled participants who completed testing for the study; time taken to complete testing
Attendance | Immediately after the intervention
  Proportion of participants who attend at least 6 of 8 scheduled Zoom visits
Completion of home practice log | Immediately after the intervention
  Proportion of of participants who complete the home practice log each week
Participant satisfaction | Immediately after the intervention
  Participant satisfaction with program, visual analog scale from 1 to 10 (10 indicating highest satisfaction)
Proportion lost to follow-up | Immediately after the intervention
  Proportion of enrolled participants who were lost to follow-up (unable to be contacted during study)

SECONDARY OUTCOMES:
Frailty index | Baseline and immediately after the intervention
  Measurement of a frailty index based on the deficit accumulation model (PMID: 32072368)
Loneliness | Baseline and immediately after the intervention
  University of California at Los Angeles 3-item Loneliness Questionnaire
Self-reported health | Baseline and immediately after the intervention
  General health perception (from SF-12)
Godin Leisure-Time Exercise Questionnaire | Baseline and immediately after the intervention
  Physical activity
Self-efficacy | Baseline and immediately after the intervention
  1 question from New General Self-Efficacy Scale
Patient health questionnaire 2-item scale (PHQ-2) | Baseline and immediately after the intervention
  Depression
Generalized Anxiety Disorder 2-item scale (GAD-2) | Baseline and immediately after the intervention
  Anxiety
Sleep | Baseline and immediately after the intervention
  Sleep questions from Patient Reported Outcome Measurement Information System (PROMIS-29) questionnaire
Short Physical Performance Battery (SPPB) | Baseline and immediately after the intervention
  Measures of balance, gait speed, and chair stands

CONTACTS AND LOCATIONS:
Overall Officials: Julia Loewenthal, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States